CLINICAL TRIAL: NCT05815277
Title: Awareness of Emergency Management of Permanent Teeth Avulsion in Children Among a Group of Egyptian Parents: a Cross Sectional Study.
Brief Title: Awareness of Parents About Management of Dental Avulsion
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Enas Abdelbadea Abdelghani Hassan, principle investigator, Cairo University
Other Study IDs: PEDO 1-1-1
Record Dates: First submitted 2023-04-02; First posted 2023-04-18 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Dental Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parents who have children aged from 6 to 12 years

SUMMARY:
Aim of the study:

assessment of level of awareness of parents about emergency management of permanent teeth avulsion in children

DETAILED DESCRIPTION:
our study asses level by awareness of parents about emergency management of dental avulsion through questionnaire , the study will be done in diagnosis clinic of faculty of oral and dental medicine Cairo university

ELIGIBILITY:
Inclusion Criteria:

* parents who have children aged from 6 to 12 years

Exclusion Criteria:

* parents who refused to participate in questionnaire
* parents who have children above or below this age

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: the patients going to diagnostic clinic of pediatric dentistry and dental public health department, Cairo university
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
level of awareness of parents about emergency management of avulsed permanent teeth | 2 months
  outcome will be assessed through a questionnaire that include binary and multiple choice questions

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine Cairo University, Cairo, Egypt